CLINICAL TRIAL: NCT04809519
Title: Effect of Integrative Nursing Based Multimodal Interventions on Blood Pressure, Stress and Treatment Compliance Levels in Uncontrolled Hypertensives: Randomized Controlled Trial
Brief Title: Integrative Nursing Based Multimodal Interventions for Uncontrolled Hypertensives
Acronym: UHTINuM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayse Dagistan Akgoz, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0030
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Uncontrolled Hypertension; Treatment Compliance; Behavior, Health; Nurse's Role
Keywords: Uncontrolled Hypertension; Treatment Adherence and Compliance; Integrative Medicine; Holistic Nursing; Yoga; Meditation; Breathing Exercises; Blood Pressure; Blood Pressure Monitoring, Home; Blood Pressure Monitoring, Self
MeSH Terms: conditions — Patient Compliance; Health Behavior; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UHTINuM (Experimental): UHTINuM is an acronym that defines multimodal interventions consisting of three components. These interventions are as follows: (1) Structured yoga program including meditation and breathing techniques (2) Hypertensive Treatment Compliance Training (3) Teaching blood pressure measurement and monitoring at home.
  Interventions: Other: Integrative Nursing based Multimodal Interventions for Uncontrolled Hypertensives
- Control group (Active Comparator): Control group will be receive information notes and standard brochures related to physical activity, healthy lifestyle behaviors advice, stop smoking etc. and will be referred to a specialist physician.
  Interventions: Other: Ongoing treatment

INTERVENTIONS:
Other: Integrative Nursing based Multimodal Interventions for Uncontrolled Hypertensives — In this study, multimodal interventions including yoga, meditation, and breathing techniques, compliance training for hypertension treatment, and home blood pressure measurement training will be applied to the experimental group.
  Arms: UHTINuM
Other: Ongoing treatment — The ongoing health service of the control group will continue. In addition, the control group will be directed to a specialist doctor and standard brochures prepared by the Ministry of Health for hypertensive individuals will be given.
  Arms: Control group

SUMMARY:
Purpose: The aim of this study is to evaluate the effect of multimodal interventions based on Integrative Nursing (IN) principles on blood pressure, stress, and hypertensive treatment compliance levels in individuals living in the community and with uncontrolled hypertension.

Design: This is a single-center, 1:1 randomized, single-blind, parallel, active comparator trial.

Method: Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) Statement 2013 checklist is used in this study. In the study, the group in which Integrative Nursing Principles-Based Multimodal Interventions were applied (UHTINuM) was taken as the experimental (n: 24), the group in which health recommendations were given as the active comparator group (n: 24). The sample size calculated according to the reference study data is 62. However, this target number could not be reached due to the COVID-19 pandemic conditions. This study was carried out with adult individuals aged 50-65 in Hayat Park, which is located within the borders of Konyaaltı District of Antalya province. Multimodal interventions including 12-week meditation and breathing techniques, yoga, hypertension treatment compliance training, and home blood pressure measurement training were applied to the UHTINuM group. The control group was directed to a specialist doctor as an intervention, information notes for hypertensive individuals and standard brochures prepared by the Ministry of Health were given. The primary results of the study were measured using an aneroid and automatic blood pressure device (blood pressure measurement), Hill Bone Hypertension Treatment Adherence Scale, Perceived Stress Scale (PSS).

This will be the first study to evaluate the effect of multimodal interventions based on integrative nursing principles in uncontrolled hypertensives. If the hypotheses of the study are reached, it is expected that the planned intervention protocol will be used by other researchers and thus become widespread in the literature. Also, the results will help contribute to the provision of care in terms of IN.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with hypertension and using regular medication for at least 1 year
* Despite being diagnosed with hypertension, systolic blood pressure 140-159 diastolic blood pressure exceeding 90-99 mmHg
* Being between the ages of 50-65
* Not being an obstacle to physical activity
* Volunteering to participate in research

Exclusion Criteria:

* The individual is not at a cognitive level to answer the questions asked.
* Having a mental illness that prevents the individual from participating in the initiative according to his / her own declaration.
* Stage 2 hypertension (SBP> 160 mm Hg or diastolic blood pressure ≥100 mm Hg)
* Having a renal problem and cardiovascular disease in which activity is prohibited by the specialist physician according to the statement of the individual.
* BMI> 40
* Having practiced yoga once a month in the last 6 months Serious musculoskeletal problems such as spinal stenosis, which, according to the individual's statement, may limit participation in yoga.
* The individual is using other mind-body therapies such as Qigong, tai chi or meditation.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | For 12 weeks
  Official and self-Blood Pressure Measurements
Perceived Stress Level | For 12 weeks
  Perceived Stress Scale: A minimum of 0 and a maximum of 32 points are obtained from the scale. Higher total score means higher perceived stress level.
Hypertensive Treatment Compliance | Change from Baseline Hypertensive Treatment Compliance at 12 months
  Hill-Bone Compliance to High Blood Pressure Therapy Scale: The scale total score varies between 0 and 42 in relation to the number of items. The scores are evaluated for the interpretation of the total, medical, nutrition and interview sub-dimension compliance scores of the scale; If the person gets "0" points in total by giving the most positive answers to all questions, he / she is considered to be fully compatible.

SECONDARY OUTCOMES:
Physical activity level | Change from Baseline Physical activity level at 12 months
  International Physical Activity Questionnaire: The short form (seven questions) obtains information about walking, moderate and intense activities, and time spent sitting. The energy required for the activities is calculated by the MET minute score. The score obtained is classified as nonphysical (MET ≤ 600 energy level), insufficient physical activity level (MET = 600-3000 energy level), and sufficient physical activity level (MET ≥3000 energy level).
BMI | Change from Baseline BMI at 12 months
  height and weight measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Community Social Area (Hayat Park), Antalya, Konyaaltı, Turkey (Türkiye)

REFERENCES:
- [Derived] Dagistan Akgoz A, Gozum S. Integrative, multimodal nursing intervention for uncontrolled hypertension: randomized controlled trial effects on blood pressure, perceived stress, and medication adherence. Clin Hypertens. 2026 Feb 1;32:e6. doi: 10.5646/ch.2026.32.e6. eCollection 2026. PMID 41660670